CLINICAL TRIAL: NCT06266611
Title: Cannabis for Palliative Care in Cancer: A Placebo-controlled Randomized Trial of Full Spectrum Hemp-derived CBD/THC
Brief Title: Cannabis for Palliative Care in Cancer
Acronym: ARCTiC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-0982
Record Dates: First submitted 2024-01-23; First posted 2024-02-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Sleep; Anxiety; Depression; Pain
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Full-Spectrum Hemp-Derived CBD (fsCBD) (Experimental): 8 weeks of use of a daily dose of cannabis (200mg CBD/4mg THC)
  Interventions: Drug: fsCBD Cannabidiol
- Broad-Spectrum Hemp-Derived CBD (bsCBD) (Experimental): 8 weeks of use of a daily dose of cannabis (200mg CBD)
  Interventions: Drug: bsCBD Cannabidiol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fsCBD Cannabidiol — Full Spectrum hemp-derived CBD (fsCBD; 200mg CBD/4mg THC) capsules produced by Ecofibre/Ananda Hemp will be used
  Arms: Full-Spectrum Hemp-Derived CBD (fsCBD)
Drug: Placebo — Placebo arm; capsules produced by Ecofibre/Ananda Hemp will be used
  Arms: Placebo
Drug: bsCBD Cannabidiol — Broad spectrum hemp-derived CBD (bsCBD; 200mg CBD) capsules produced by Ecofibre/Ananda Hemp will be used
  Arms: Broad-Spectrum Hemp-Derived CBD (bsCBD)

SUMMARY:
Many cancer patients suffer from pain, sleep, and mood problems and are using cannabis to relieve these symptoms. Cannabis may provide such relief but may also produce negative side effects including cognitive impairment, an especially problematic issue for cancer patients, indicating more research on cannabis use in the cancer context is required. In this endeavor, the present study seeks to compare the use of hemp-derived CBD (Cannabidiol) with and without THC (Delta-9-tetrahydrocannabinol) versus placebo on measures of sleep, pain, mood, subjective and objective cognitive functioning, and quality of life within 185 cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Aged ≥25 years at Visit 1 (Baseline)
3. Have a diagnosis of any solid tumor type and is currently undergoing or has undergone either curative or palliative treatment in the past 18 months
4. Currently experiencing symptoms of sleep problems, pain, and/or mood disturbance (i.e., depression, anxiety)
5. Desire to use cannabis to treat their symptoms
6. Must not have been regularly using any cannabis products (more than 3x/month) in the last 6 months
7. Willing to practice acceptable methods of birth control until completing study medication

Exclusion Criteria:

1. Report of illegal drug use (e.g., cocaine, methamphetamine) in the past 90 days
2. Current use of anti-epileptic medications (e.g., clobazam, sodium valproate, lamotrigine)
3. Current use of medications known to have major interactions with Epidiolex (e.g., buprenorphine, leflunomide, levomethadyl acetate, lomitapide, mipomersen, pexidartinib, propoxyphene, sodium oxybate, teriflunomide)
4. Current use of anti-psychotic medications
5. Current use of potent CYP2C19 or CYP3A4 inducers (e.g., Rifampin, apalutamide, carbamazepine, enzalutamide, ivosidenib9, lumacaftor, ivacaftor, phenytoin, St. John's wort, Fosphenytoin, Mitotane, Phenobarbital, Primidone)
6. Liver function tests (Alanine transaminase [ALT] and Aspartate transaminase [AST]) levels ≥2x the upper normal limits
7. Moderate or severe liver disease
8. Past or current diagnosis, or family history of diagnosis, of psychosis; current major psychiatric illness, such as bipolar disorder, major depression, or schizophrenia
9. History of seizures
10. For female participant of childbearing potential: Pregnant or lactating at the time of study enrollment or trying to become pregnant. Lack of childbearing potential confirmed by a history of amenorrhea for at least 12 consecutive months and serum FSH level within the laboratory's reference range for postmenopausal females OR documented bilateral oophorectomy and/or hysterectomy
11. Physician response to passive consent indicating contraindications for participation.
12. Unwilling to refrain from cannabis use other than study drug for the entire study duration
13. Men who consume more than 2 alcoholic beverages per day and women who consume more than 1 alcoholic beverage per day

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Interference | Baseline, 4 weeks, 8 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference. Total scores are between 8 and 40, with higher scores meaning more pain interference.
Pain Intensity | Baseline, 4 weeks, 8 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Intensity (7-day). Scores are between 0-10, with 0 being no pain and 10 being the worst imaginable pain.
Pain Inventory | Baseline, 4 weeks, 8 weeks
  Brief Pain Inventory (BPI) survey. Measures pain levels, pain interference, and relief from medication, and includes diagrams for labeling pain. For pain levels, various questions ask participants to rate pain on a scale of 0-10, 0 being no pain and 10 being pain as bad as you can imagine. For questions about pain interference, each question is on a scale of 0-10, where 0 does not interfere and 10 completely interferes. BPI is scored as an average of each subsection, where a higher average suggests greater severity of pain/more interference.
Sleep Disturbance | Baseline, 4 weeks, 8 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disturbance 4a. Scores are separated between the first question (sleep quality) and the remaining 7 questions. For the first question, scores are between 1 and 5, with 1 being very poor sleep quality and 5 being very good sleep quality. The remaining 7 questions are scored individually on a scale of 1--5; for some questions, higher scores mean less disturbance, and for others, a higher score means more disturbance.
Sleep-Related Impairment | Baseline, 4 weeks, 8 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep-Related Impairment 4a. Scores are between 4 and 20, with higher scores indicating more sleep-related impairment
Depression/Anxiety | Baseline, 4 weeks, 8 weeks
  Depression Anxiety Stress Scale - 21 Item (DASS-21). Scores are between 0 and 63, with higher scores indicating more negative emotional states.
Fatigue | Baseline, 4 weeks, 8 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Fatigue 4a. Scores range from 4-20, with higher scores indicating more fatigue.
Health Related Quality of Life | Baseline, 4 weeks, 8 weeks
  Health Related Quality of Life Short Form 12 (SF-12). Scores range from 0-100 with higher scores indicating better health.
FACT-Cog Cognitive Function | Baseline, 4 weeks, 8 weeks
  Functional Assessment of Cognitive Function - Cognitive (FACT-Cog). Scores are transformed such that scores range from 0-132 and higher scores indicate a better quality of life/cognitive function.
Stroop Task Test of Cognitive Function | Baseline, 4 weeks, 8 weeks
  Stroop Task
DSST Test of Cognitive Function | Baseline, 4 weeks, 8 weeks
  Digit Symbol Substitution Task (DSST)
Conners Test of Cognitive Function | Baseline, 4 weeks, 8 weeks
  Conners Continuous Performance Test - Version 3 (CPT-3)
Plasma Cannabinoids | Baseline, 4 weeks, 8 weeks
  Plasma cannabinoid levels in participants will be measured from biological samples.
PROMIS Pain Intensity (Right Now) | 4 weeks
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Intensity (Right Now). Scores are between 0-10, with 0 being no pain and 10 being the worst imaginable pain.
Drug Effects | 4 weeks
  Drug Effects Questionnaire (DEQ). Six questions about drug effects with possible answers of "not at all", "somewhat", and "extremely", where higher scores indicate higher drug effects.
ARCI-Marijuana Scale | 4 weeks
  Addiction Research Center Inventory - Marijuana Scale (ARCI-M). 12 True or false questions where more "true" answers indicate higher drug effects.
Drug Effects - Mood | 4 weeks
  Profile of Mood States (POMS). Scores are between 28-140, with higher scores indicating higher drug effects.
Drug Effects - Blood Cannabinoids | 4 weeks
  Acute plasma cannabinoid levels in participants will be measured from blood samples pre-drug administration, on-hour post drug administration, and 2-hours post drug administration at week 4 appointment.

SECONDARY OUTCOMES:
Polypharmacy for Pain | Baseline, 4 weeks, 8 weeks
  Use of pain medications
Polypharmacy for Psychiatric Rx | Baseline, 4 weeks, 8 weeks
  Use of psychiatric medications
Polypharmacy for Sleep | Baseline, 4 weeks, 8 weeks
  Use of sleep medications

OTHER OUTCOMES:
Cancer Treatment Type | Baseline
  Type of treatment participant is using for cancer, including specific type of immunotherapy, if relevant and known
Cancer Disease Progression | Baseline, 4 weeks, 8 weeks
  Assess cancer disease progression and report as outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Anschutz Health Sciences Building, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No